CLINICAL TRIAL: NCT03373942
Title: Evaluation of Choroidal Thickness Using Spectral Optical Coherence Tomography in Pseudoexfoliation Glaucoma and Primary Open Angle Glaucoma
Brief Title: The Effect of Pseudoexfoliation on Choroidal Thickness in Open Angle Glaucoma
Status: Completed | Type: Observational
Sponsor: Emine Deniz Egrilmez (Other)
Collaborators: Izmir Ataturk Training and Research Hospital (Other)
Responsible Party: Sponsor-Investigator, Emine Deniz Egrilmez, M.D., Izmir Ataturk Training and Research Hospital
Organization: Izmir Ataturk Training and Research Hospital (Other)
Other Study IDs: 256/30.12.2015
Record Dates: First submitted 2017-11-06; First posted 2017-12-14 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Glaucoma, Open-Angle
Keywords: glaucoma; EDI OCT; pseudoexfoliation; choroidal thickness
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary Open Angle Glaucoma (POAG): The study included 30 eyes of 30 patients diagnosed with POAG who presented to Glaucoma Unit of İzmir Katip Çelebi University Atatürk Training and Research Hospital
  Interventions: Other: Choroidal thickness measurements with SD-OCT device
- Pseudoexfoliation Syndrome (PEX): The study included 30 eyes of 30 patients diagnosed with PEX glaucoma who presented to Glaucoma Unit of İzmir Katip Çelebi University Atatürk Training and Research Hospital
  Interventions: Other: Choroidal thickness measurements with SD-OCT device
- Control: The control group included 30 eyes of 30 healthy individuals with similar age distribution with POAG and PEX group
  Interventions: Other: Choroidal thickness measurements with SD-OCT device

INTERVENTIONS:
Other: Choroidal thickness measurements with SD-OCT device
  Other Names: General ophthalmological examination; Visual field examination; Optical biometry

SUMMARY:
Purpose: To investigate the effect of pseudoexfoliation (PEX) on choroidal thickness in primary open-angle glaucoma (POAG).

Methods: This prospective, randomized study included 30 POAG patients and 30 PEX glaucoma patients with similar demographic characteristics, and 30 eyes of 30 healthy individuals comprised the control group. Macular choroidal thickness was measured using a Cirrus HD spectral domain optical coherence tomography (OCT) instrument.

DETAILED DESCRIPTION:
In the present study, the investigators aimed to evaluate the effect of the presence of PEX on choroidal thickness in two groups of glaucoma patients with similar degrees of damage and similar demographical characteristics. The investigators also evaluated whether there was a correlation between choroidal thickness and indicators of glaucoma severity, such as retinal nerve fiber layer (RNFL) thickness and mean deviation (MD) value, in these two glaucoma types.

MATERIALS AND METHODS The study included 30 eyes of 30 patients diagnosed with POAG and 30 eyes of 30 patients diagnosed with PEX glaucoma who presented to Glaucoma Unit of Izmir Katip Celebi University Atatürk Training and Research Hospital between August 2014 and February 2015. The control group included 30 eyes of 30 healthy individuals with similar age distribution.

Approval was obtained from the ethics committee of Izmir Katip Celebi University Medical School Atatürk Training and Research Hospital. Detailed informed consent forms were obtained from each of the patients included in the study.

The study included subjects over 18 years old who had best corrected visual acuity of 0.5 or better, transparent optic medium, at least two reliable visual field tests, and reliable spectral domain (SD)-OCT (signal strength≥7/10) and EDI-OCT images (signal strength≥6/10) Information pertaining to patients' systemic diseases and chronic medication use was recorded. Patients with diabetes mellitus, systemic arterial hypertension, renal failure, hemodialysis history, chronic medication, or smoking habit were not included.

Patients with retinal and neuro-ophthalmological diseases, amblyopia, active or previous uveitis, previous ocular trauma, intraocular surgery within last 6 months, previous trabeculectomy, or refractive error with a spherical equivalent greater than ±3.0 D were excluded from the study. In order to minimize the effect of IOP on choroidal thickness, patients with IOP higher than 21 mmHg at the time of OCT image acquisition were not included in the study.

POAG was diagnosed based on high IOP (>21 mmHg) at the time of diagnosis, typical glaucomatous optic disc and visual field changes, and normal anterior chamber angle. In contrast, PEX glaucoma diagnosis was based on high IOP (>21 mmHg) at diagnosis and typical glaucomatous optic disc and visual field changes, plus the presence of PEX material or hyperpigmentation in the anterior chamber angle and the presence of PEX material at the pupillary margins or the anterior lens on anterior segment examination after pupil dilation. The control group consisted of healthy individuals with normal anterior and posterior segment findings and IOP less than 21 mmHg.

All subjects underwent a detailed ophthalmologic examination. Axial length was measured using IOL Master (Carl Zeiss Meditec, Dublin, CA, USA) optic biometry. Visual field was assessed with Humphrey II Perimetry (Carl Zeiss Meditec, Dublin, CA, USA) SITA standard central 24-2 test. Tests with fixation loss less than 20%, false negative, and false positive response rates below 33% were considered reliable. Patients with at least two reliable visual field tests were included in the study. MD values were obtained.

Optic disc images were obtained with Cirrus 4000 HD-OCT (Carl ZeissMeditec, Dublin, CA, USA) SD-OCT device. Mean RNFL thickness and vertical cup-to-disc (c/d) ratios were noted. Choroidal imaging was done after pupil dilation using the EDI-OCT mode. The SD Cirrus HD-OCT light source was centered on 800 nm wavelength to achieve 5 μm maximal resolution in tissue. In order to minimize the effect of diurnal choroidal thickness variation on the measurements, choroidal thickness measurements of all patients were made between 09:00 and 11:00 am, after a resting period of 30 minutes. The macular field was scanned in the horizontal plane in high-resolution 1 line raster mode. Patients were asked to focus on the instrument's internal fixation light until the retinal image was acquired. Images with signal strength of 6/10 or better were eligible for assessment. Patients who had at least two reliable high-resolution foveal and choroidal imagings were included in the study.

The fovea centralis was determined by identifying the point of maximum depression in the central 500-micron-diameter area. The internal and external choroidal margins were determined manually in the section passing through the fovea centralis. These margins were drawn based on criteria defined by Boonarpha et al.[15]. The posterior edge of the hyperreflective band corresponding to the retinal pigment epithelium-Bruch's membrane complex was determined as the anterior border of the choriocapillaris. The posterior border of the choriocapillaris was demarcated as the hyperreflective band corresponding to the sclerochoroidal interface or the hyporeflective line corresponding to suprachoroidal space. In cases where these two anatomic structures could not be visualized, measurement was done using the prominent straight line corresponding to the posterior margin of the large choroidal vessels. Patients in whom choroidal margins could not be clearly distinguished were not included in the study.

High-resolution retinal choroidal images with distinct choroidal margins were transferred to ImageJ software [40]. The high-resolution EDI-OCT images were 6000 microns wide and 2000 microns high, as indicated in the manufacturer's user's manual. EDI-OCT images to be measured were opened using ImageJ software. The Scale command was selected in the Image tab of ImageJ software menu. Using the Scale menu, width (pixels) was defined as 6000 and height (pixels) as 2000. The distance to be measured was marked on the new image of 6000x2000 pixels and measurements were done using the Measure command in Analyze tab. The choroidal margins were drawn in this software according to the specified criteria, followed by manual measurements. Measurements were taken vertically at the fovea centralis and in the nasal and temporal quadrants at distances of 1500 and 2500 microns from the fovea centralis. The same researcher repeated the measurements at different times using the double-blind method, and intraobserver and intervisit measurement repeatability was assessed.

All data were analysed using SPSS software. Independent t-test was used to compare the groups. The correlation between choroidal thickness and other variables (age, axial length, vertical c/d, RNFL thickness, MD) was evaluated using Pearson correlation analysis.Repeatability analysis of study parameters measured with Cirrus 4000 HD OCT was evaluated using the coefficient of variation (CV). For CV calculation of choroidal thickness measured by Cirrus 4000 HD OCT, 10 consequential measurements were obtained by the same operator to the same eye of the subject. CV is defined as the ratio of the standard deviation to the mean: cV=σ/μ

ELIGIBILITY:
Inclusion Criteria:

* The study included subjects over 18 years old who had best corrected visual acuity of 0.5 or better, transparent optic medium, at least two reliable visual field tests, and reliable spectral domain (SD)-OCT (signal strength≥7/10) and EDI-OCT images (signal strength≥6/10)

Exclusion Criteria:

* Information pertaining to patients' systemic diseases and chronic medication use was recorded. Patients with diabetes mellitus, systemic arterial hypertension, renal failure, hemodialysis history, chronic medication, or smoking habit were not included.
* Patients with retinal and neuro-ophthalmological diseases, amblyopia, active or previous uveitis, previous ocular trauma, intraocular surgery within last 6 months, previous trabeculectomy, or refractive error with a spherical equivalent greater than ±3.0 D were excluded from the study. In order to minimize the effect of IOP on choroidal thickness, patients with IOP higher than 21 mmHg at the time of OCT image acquisition were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: POAG was diagnosed based on high IOP (>21 mmHg) at the time of diagnosis, typical glaucomatous optic disc and visual field changes, and normal anterior chamber angle. In contrast, PEX glaucoma diagnosis was based on high IOP (>21 mmHg) at diagnosis and typical glaucomatous optic disc and visual field changes, plus the presence of PEX material or hyperpigmentation in the anterior chamber angle and the presence of PEX material at the pupillary margins or the anterior lens on anterior segment examination after pupil dilation. The control group consisted of healthy individuals with normal anterior and posterior segment findings and IOP less than 21 mmHg.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-08-15 (Actual); Primary Completion 2015-02-15 (Actual); Study Completion 2015-08-15 (Actual)

PRIMARY OUTCOMES:
The Effect of Pseudoexfoliation on Choroidal Thickness in Open Angle Glaucoma | Between August 2014 and February 2015
  Choroidal thicknesses at nasal 2500 µm, nasal 1500 µm, subfoveal, temporal 1500 µm, and temporal 2500 µm in the three groups were measured

CONTACTS AND LOCATIONS:
Overall Officials: Seyda K Ugurlu, Prof, Study Director — Izmir Katip Celebi University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anastasopoulos E, Founti P, Topouzis F. Update on pseudoexfoliation syndrome pathogenesis and associations with intraocular pressure, glaucoma and systemic diseases. Curr Opin Ophthalmol. 2015 Mar;26(2):82-9. doi: 10.1097/ICU.0000000000000132. PMID 25594764
- [Background] Andrikopoulos GK, Alexopoulos DK, Gartaganis SP. Pseudoexfoliation syndrome and cardiovascular diseases. World J Cardiol. 2014 Aug 26;6(8):847-54. doi: 10.4330/wjc.v6.i8.847. PMID 25228963
- [Background] Ritch R, Schlotzer-Schrehardt U. Exfoliation syndrome. Surv Ophthalmol. 2001 Jan-Feb;45(4):265-315. doi: 10.1016/s0039-6257(00)00196-x. PMID 11166342
- [Background] Konstas AG, Stewart WC, Stroman GA, Sine CS. Clinical presentation and initial treatment patterns in patients with exfoliation glaucoma versus primary open-angle glaucoma. Ophthalmic Surg Lasers. 1997 Feb;28(2):111-7. PMID 9054481
- [Background] Manjunath V, Taha M, Fujimoto JG, Duker JS. Choroidal thickness in normal eyes measured using Cirrus HD optical coherence tomography. Am J Ophthalmol. 2010 Sep;150(3):325-329.e1. doi: 10.1016/j.ajo.2010.04.018. Epub 2010 Jun 29. PMID 20591395
- [Background] Margolis R, Spaide RF. A pilot study of enhanced depth imaging optical coherence tomography of the choroid in normal eyes. Am J Ophthalmol. 2009 May;147(5):811-5. doi: 10.1016/j.ajo.2008.12.008. Epub 2009 Feb 20. PMID 19232559
- [Result] Zhang Z, Yu M, Wang F, Dai Y, Wu Z. Choroidal Thickness and Open-Angle Glaucoma: A Meta-Analysis and Systematic Review. J Glaucoma. 2016 May;25(5):e446-54. doi: 10.1097/IJG.0000000000000275. PMID 25943737
- [Result] Bayhan HA, Bayhan SA, Can I. Evaluation of the Macular Choroidal Thickness Using Spectral Optical Coherence Tomography in Pseudoexfoliation Glaucoma. J Glaucoma. 2016 Feb;25(2):184-7. doi: 10.1097/IJG.0000000000000100. PMID 25122536
- [Result] Zengin MO, Cinar E, Karahan E, Tuncer I, Yilmaz S, Kocaturk T, Kucukerdonmez C. Choroidal thickness changes in patients with pseudoexfoliation syndrome. Int Ophthalmol. 2015 Aug;35(4):513-7. doi: 10.1007/s10792-014-9977-x. Epub 2014 Jul 25. PMID 25059402
- [Result] Goktas S, Sakarya Y, Ozcimen M, Sakarya R, Bukus A, Ivacik IS, Erdogan E. Choroidal thinning in pseudoexfoliation syndrome detected by enhanced depth imaging optical coherence tomography. Eur J Ophthalmol. 2014 Nov-Dec;24(6):879-84. doi: 10.5301/ejo.5000460. Epub 2014 Apr 4. PMID 24729143
- [Result] Eroglu FC, Asena L, Simsek C, Kal A, Yilmaz G. Evaluation of choroidal thickness using enhanced depth imaging by spectral-domain optical coherence tomography in patients with pseudoexfoliation syndrome. Eye (Lond). 2015 Jun;29(6):791-6. doi: 10.1038/eye.2015.34. Epub 2015 Mar 27. PMID 25853396
- [Result] Ozge G, Koylu MT, Mumcuoglu T, Gundogan FC, Ozgonul C, Ayyildiz O, Kucukevcilioglu M. Evaluation of retinal nerve fiber layer thickness and choroidal thickness in pseudoexfoliative glaucoma and pseudoexfoliative syndrome. Postgrad Med. 2016 May;128(4):444-8. doi: 10.1080/00325481.2016.1170579. Epub 2016 Apr 4. PMID 27007173
- [Result] Turan-Vural E, Yenerel N, Okutucu M, Yildiz E, Dikmen N. Measurement of Subfoveal Choroidal Thickness in Pseudoexfoliation Syndrome Using Enhanced Depth Imaging Optical Coherence Tomography. Ophthalmologica. 2015;233(3-4):204-8. doi: 10.1159/000371899. Epub 2015 Feb 7. PMID 25676024
- [Result] Kocabeyoglu S, Uzun S, Kadayifcilar S, Mocan MC, Irkec M. The Relationship Between Choroidal Expansion and Intraocular Pressure Rise During the Water Drinking Test in Healthy Subjects and Patients With Exfoliation Syndrome. J Glaucoma. 2016 Apr;25(4):e324-8. doi: 10.1097/IJG.0000000000000283. PMID 26035419
- [Result] Demircan S, Yilmaz U, Kucuk E, Ulusoy MD, Atas M, Gulhan A, Zararsiz G. The Effect of Pseudoexfoliation Syndrome on the Retinal Nerve Fiber Layer and Choroid Thickness. Semin Ophthalmol. 2017;32(3):341-347. doi: 10.3109/08820538.2015.1090611. Epub 2016 Apr 14. PMID 27077400
- [Result] Mwanza JC, Hochberg JT, Banitt MR, Feuer WJ, Budenz DL. Lack of association between glaucoma and macular choroidal thickness measured with enhanced depth-imaging optical coherence tomography. Invest Ophthalmol Vis Sci. 2011 May 18;52(6):3430-5. doi: 10.1167/iovs.10-6600. PMID 21357398